CLINICAL TRIAL: NCT01373749
Title: Compare of Continued Nitro Oxide Inhalation and Nitro Oxide Inhalation Continued With Oral Sildenafil on Treatment of Neonatal Persistent Pulmonary Hypertension
Brief Title: Nitro Oxide Inhalation Continued With Sildenafil on Neonatal Persistent Pulmonary Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Military Medical University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Dr.Hu.Zhangxue, Department of Pediatrics, Daping Hospital, Third Military Medical Universityof PLA,CHINA
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1991660
Record Dates: First submitted 2011-05-31; First posted 2011-06-15 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2011-01

CONDITIONS: Persistent Pulmonary Hypertension of Newborn
Keywords: PPHN; NO inhalation; Sildenafil; Treatment; Safety
MeSH Terms: conditions — Persistent Fetal Circulation Syndrome | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NOS (Experimental): NO inhalation was performed in the first stage(<48h) of PPHN, NO inhalation was replaced by sildenafil in the second stage(>48h).
  Interventions: Drug: NO inhalation continued with sildenafil
- NO (Placebo Comparator): NO inhalation was performed during the whole treatment procedure of PPHN. There is no other methods given to treat PPHN during the therapy course.
  Interventions: Drug: NO inhalation

INTERVENTIONS:
Drug: NO inhalation — NO inhalation was performed as the only treatment for PPHN during the whole course.
  Arms: NO
Drug: NO inhalation continued with sildenafil — NO inhalation was performed as the primary treatment for PPHN in the first 48 hours, NO inhalation will be replaced by sildenafil after 48 hours of therapy.
  Arms: NOS

SUMMARY:
Nitro Oxide (NO) inhalation was recognized as an effect treatment of Neonatal Persistent Pulmonary Hypertension (PPHN), while the safety of NO long term application was under investigation. Several research suggested too much NO2 was generated in the lung after long term (> 72h) use of NO inhalation, which cause bad effects on PS production.

Sildenafil was proved to be effective to PPHN as NO. This medication has a similar clinical effect but need monitoring of blood pressure. The possible hypotension effect restrict the dosage of sildenafil, which limit the usage of sildenafil in severe PPHN. But we recommend sildenafil to The purpose of the study was to establish if NO continued with sildenafil has the same effect as single NO inhalation.

ELIGIBILITY:
Inclusion Criteria:Diagnosed as PPHN in the NICU,primary disease:neonate respiratory distress syndrome,meconium aspiration syndrome of newborn,severe neonatal infectious pneumonia.

* Pulmonary artery pressure > 50mmHg
* mechanical ventilation over 48h
* primary OI(PO2/FiO2)<300
* difference of SpO2 between up and low limbs > 10%
* high FiO2 oxygen inhalation test: positive

Exclusion Criteria:

* congenital heart disease
* diaphragmatic hernia

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-12 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
persistent normal pulmonary artery pressure | 96 hours
  The pulmonary artery pressure returned back to a normal level(<30mmHg) and last over 48 hours.

SECONDARY OUTCOMES:
Recover without complication | 1 month after therapy
  To ensure the safety of the therapies, brain and lung complications of the baby after PPHN is going to be observed 1 month after birth.
  1. incidence of pulmonary disease;(chronic lung disease)
  2. incidence of brain injury. (Hypoxic-ischemic encephalopathy)
  3. Heart structure change(right ventricle enlarge)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatrics,Daping hospital, Chongqing, Chongqing Municipality, China